CLINICAL TRIAL: NCT01854489
Title: Effects of Rifampicin on the Pharmacokinetics and Pharmacodynamics of Sublingual and Intravenous Buprenorphine: A Four-phase Cross-over Study in Healthy Subjects.
Brief Title: Effects of Rifampicin on the Pharmacokinetics and Pharmacodynamics of Sublingual and Intravenous Buprenorphine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Mari Fihlman, MD, Turku University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Rifabupre
Record Dates: First submitted 2013-04-27; First posted 2013-05-15 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Buprenorphine; Rifampicin; Interactions; Pharmakokinetics; Pharmakodynamics
MeSH Terms: interventions — Rifampin; Buprenorphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rifampicin (Active Comparator): The volunteers will be given oral rifampicin (Rimapen, Orion, Finland) 600 mg as a single daily dose at 20.00 for 7 days
  Interventions: Drug: Rifampicin
- Placebo (Placebo Comparator): The volunteers will be given oral placebo at 20.00 for 7 days
  Interventions: Drug: Placebo
- Buprenorphine (Active Comparator): The volunteers will be given single dose of 0,4 mg intra venous buprenorphine or 0,6 mg sublingual buprenorphine on day 5.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Placebo — The volunteers will be given Oral placebo at 20.00 for 7 days [Phase 1 ]
  Arms: Placebo
Drug: Rifampicin — The volunteers will be given oral rifampicin (Rimapen, Orion, Finland) 600 mg as a single daily dose at 20.00 for 7 days
  Arms: Rifampicin
Drug: Buprenorphine — The volunteers will be given single dose of 0,4 mg intra venous buprenorphine or 0,6 mg sublingual buprenorphine on day 5.
  Other Names: Temgesic 0,2 mg resoriblet; Temgesic 0,3 mg/ml
  Arms: Buprenorphine

SUMMARY:
This study is aimed to examine the possible interactions of sublingual and intravenous buprenorphine with rifampicin.

DETAILED DESCRIPTION:
Variability in drug response can be due to either pharmacokinetic or pharmacodynamic factors. The reasons why people differ in pharmacokinetics or pharmacodynamics are manifold and include, e.g., genetic factors, diseases, age and concomitantly administered drugs. Oxidation reactions are dominant in the metabolism of drugs and cytochrome P-450 enzymes (CYP) have been recognized as chief contributors. We have previously shown that drug interactions mediated by the inhibition of CYP enzymes may be of major clinical significance.Buprenorphine is a semisynthetic partial µ-opioid receptor agonist. In low doses, it is used in the treatment of moderate acute and chronic pain whereas in high doses, it is used in the management of opioid withdrawal symptoms and opioid addiction. It has high affinity for the µ-opioid receptor and its analgesic efficacy is 20-40 times that of morphine. It acts as an antagonist at the myy-opioid receptor and as an agonist at the myy-opioid receptor and opioid-like receptor (ORL-1).

Buprenorphine undergoes extensive first-pass metabolism and has low oral bioavailability of 15 %. Bioavailability following sublingual administration of buprenorphine is higher, 50-60 %. After high sublingual doses of buprenorphine (8-24 mg), peak plasma concentrations are reached in 1 hour and after low sublingual doses (0.4 mg) they are reached in approximately 3 h. Approximately two-thirds of a buprenorphine dose is excreted unchanged, and the rest is metabolized in the liver and intestinal wall. N-dealkylation of buprenorphine mainly via CYP3A but also CYP2C8 yields norbuprenorphine, and glucuronidation yields buprenorphine-3-glucuronide. Norbuprenorphine is excreted in the urine after subsequent conjugation. 80-90 % of buprenorphine is excreted by the biliary system and enterohepatic circulation.Although few interaction studies of high-dose buprenorphine and antiretrovirals have been conducted, the effect of CYP3A inducers on the pharmacokinetics of low-dose buprenorphine is unknown. Because the use of buprenorphine in pain management is increasing after the introduction of transdermal buprenorphin patches to the market, it is clinically relevant to study and quantify possible interactions of buprenorphine with inducers of its CYP3A-mediated metabolism such as rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* aged 18-40 years
* body weights within ±15% of the ideal weight for height

Exclusion Criteria

* A previous history of intolerance to the study drugs or to related compounds and additives.
* Concomitant drug therapy of any kind for at least 14 days prior to the study.
* Subjects younger than 18 years and older than 40 years.
* Existing or recent significant disease.
* History of hematological, endocrine, metabolic or gastrointestinal disease, including gut motility disorders.
* History of asthma or any kind of drug allergy.
* Previous or present alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements.
* A positive test result for urine toxicology.
* A "yes" answer to any one of the Abuse Questions.
* Pregnancy or nursing.
* Donation of blood for 4 weeks prior and during the study.
* Special diet or life style conditions which would compromise the conditions of the study or interpretation of the results.
* Participation in any other studies involving investigational or marketed drug products concomitantly or within one month prior to the entry into this study.
* Smoking for one month before the start of the study and during the whole study period.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Concentration of buprenorphine and its metabolites in plasma and urine concebtration of buprenorphine | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 and 20 hours after administration of buprenorphine

SECONDARY OUTCOMES:
Pharmacodynamic effects | 1, 2,3, 4, 5, 6, 8, 10, 12, 20 hours after administration of buprenorphine
  The psychomotor effects on bubrenorphine will be assessed with the measurement of pupil size, Maddox wing test and symbol substitution test.
Analgesia | 1, 2, 3, 4, 5, 6, 8, 10, 12 hours after the administration of buprenorphine
  The analgesic effect of buprenorphine will be evaluated using the cold pressor test. The cold pain test has been shown to be sensitive to opioid analgesia, and it enables repeated assessments of cold pain threshold, tolerance, intensity and unpleasantness

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland